CLINICAL TRIAL: NCT05969626
Title: A Randomized, Blinded, Parallel Controlled Phase 3 Clinical Trial to Evaluate the Immunogenicity and Safety of Freeze-dried Human Rabies Vaccine (Without Serum Vero Cells) Administered to People Aged 10-60 Years With Different Immunization Procedures
Brief Title: Clinical Trial of Freeze-dried Human Rabies Vaccine (Without Serum Vero Cells)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ningbo Rongan Biological Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AIM1813-III
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-07

CONDITIONS: Rabies
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 5-dose group of test vaccine (Experimental)
  Interventions: Biological: 5-dose group of test vaccine
- 5-dose group of control vaccine (Active Comparator)
  Interventions: Biological: 5-dose group of control vaccine
- 4-dose A group of test vaccine (Experimental)
  Interventions: Biological: 4-dose A group of test vaccine
- 4-dose B group of test vaccine (Experimental)
  Interventions: Biological: 4-dose B group of test vaccine

INTERVENTIONS:
Biological: 5-dose group of test vaccine — Subjects will be vaccinated on days 0, 3, 7, 14, and 28
  Arms: 5-dose group of test vaccine
Biological: 5-dose group of control vaccine — Subjects will be vaccinated on days 0, 3, 7, 14, and 28
  Arms: 5-dose group of control vaccine
Biological: 4-dose A group of test vaccine — Subjects will be vaccinated on days 0, 3, 7, 14
  Arms: 4-dose A group of test vaccine
Biological: 4-dose B group of test vaccine — Subjects will be vaccinated on days 0, 3, 7, 28
  Arms: 4-dose B group of test vaccine

SUMMARY:
This study was intended to explore the safety and immunogenicity of the test vaccine compared to the control vaccine. The trial consisted of two phases.

Phase I used an open-ended design. Phase II used a randomized, blinded, parallel-controlled non-inferiority design with the same type of active vaccine, in which the control vaccine 5-dose group and the test vaccine 5 group were kept blinded throughout, the test vaccine 4-dose B group was kept blinded from the other three groups until visit 4 （D14）, and the test vaccine 4-dose A group was kept blinded from the control vaccine 5-dose group and the test vaccine 5-dose group until visit 5 （D28）.

ELIGIBILITY:
Inclusion Criteria:

1. The age of the subject is 10-60 years old (≥10 years old, <61 years old);
2. Subjects aged 10-17 and their guardians can provide valid identification; subjects aged 18-60 can provide valid identification;
3. Subjects aged 10-17 and at least one of their guardians voluntarily participate with informed consent, and sign the Informed Consent for minors and adults respectively; Subjects aged 18-60 voluntarily participate with informed consent and sign the adult version of Informed Consent; Basic reading and writing skills are required;
4. If the subjects are WOCBP (women of childbearing potential), they should not be pregnant or breastfeeding, have a negative urine pregnancy test before vaccination, and have taken effective contraceptive measures within 2 weeks before being enrolled in this study; From enrollment in the study until 6 months after full exemption, no family planning and consent to use effective contraception during the study period. Effective forms of birth control include: oral contraceptives (excluding emergency contraceptives)Injectable or embedded contraception, sustained release topical contraceptives, hormonal patches, intrauterine devices, sterilization, abstinence, condoms (male), isolationMembrane, cervical cap, etc.;
5. * On the day of enrollment, armpit body temperature of subjects >14 years old was <37.3℃, and armpit body temperature of subjects <14 years old was <37.5℃;
6. Adult subjects or minor subjects and their guardians shall comply with the requirements of the clinical study protocol.

Exclusion Criteria:

* Exclusion Criteria at 1-dose:

  1. A history of rabies vaccine immunization or rabies virus passive immunization was asked;
  2. A history of grade 2 or 3 injury in animals susceptible to rabies virus (cats, dogs, etc.) within 12 months prior to the first dose of vaccination (the assessment criteria was the Technical Guidelines for Rabies Prevention and Control (2016));
  3. Plan to participate in other clinical trials during the clinical study;
  4. Allergic to any component of the test vaccine; History of severe allergies that require medical intervention, such as anaphylactic shock, allergic laryngeal edema, anaphylactoid purpura, thrombocytopenic purpura, allergic necrosis reaction (Arthus reaction), severe urticaria, dyspnea, angioneurotic edema, etc.;
  5. Have been diagnosed with a congenital or acquired immunodeficiency disease, such as HIV infection, lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease, or other immune disease that the investigator has determined may affect the evaluation of the trial;
  6. Known or suspected serious medical conditions upon inquiry include: severe respiratory diseases, poorly controlled chronic diseases, severe liver and kidney diseases, severe cardiovascular diseases, malignant tumors, etc.;
  7. * Medically unmanageable hypertension, such as systolic blood pressure >120mmHg and/or diastolic blood pressure >80mmHg in subjects 10 to 17 years of age prior to enrollment, systolic blood pressure of 140mmHg and/or diastolic blood pressure of 90mmHg in subjects 18 years of age and older;
  8. Coagulation dysfunction (e.g. coagulation factor deficiency, coagulation disorders, platelet abnormalities) or coagulation disorders diagnosed by a physician;
  9. Asplenia, functional asplenia, and any condition resulting in asplenia or splenectomy;
  10. Have received immunosuppressive therapy within 3 months prior to vaccination or plan to receive immunosuppressive therapy throughout the study period;
  11. Plan to receive such treatment within 30 days after the first dose to the full dose, such as long-term systemic glucocorticoid therapy (2 weeks or more at a dose of >2mg/kg/ day or >20mg/ day of prednisone or equivalent); Allow topical use (such as ointment, eye drops, inhalants or nasal sprays);
  12. * Received immunoglobulins or blood-related products within 3 months prior to vaccination or plan to receive them throughout the study period;
  13. * Acute illness or acute onset of chronic disease within 3 days prior to vaccination;
  14. * Antipyretic, analgesic and anti-allergic drugs were used within 3 days prior to vaccination;
  15. * Have received COVID-19 vaccine or live attenuated vaccine within 28 days prior to vaccination, and have received inactivated vaccines other than COVID-19 inactivated vaccines within 14 days prior to vaccination;
  16. Previous or current diagnosis of neurological or psychiatric disorders (including but not limited to dementia, schizophrenia, bipolar disorder, etc.) or confirmed Seizures, convulsions (excluding febrile convulsions in children 5 years of age and younger)), and other neuropsychiatric disorders deemed unsuitable for participation in this study by the investigator;
  17. Due to various medical, psychological, social, or other conditions that, in the judgment of the investigator, are inconsistent with the study protocol or cannot be complied with.

      For the criteria marked with an (*), if the subject has the conditions specified in that criteria, the visit may be rescheduled when those conditions are no longer present.

      In addition to the examination items set by the protocol, other medical history, surgical history, and medication history were obtained in the form of consultation.

      Criteria for subsequent dose delays:If any of the following conditions occur before any subsequent dose of the subject, the vaccination should be postponed until the vaccination requirements are met.

  <!-- -->

  1. On the day of vaccination, the axillary temperature is measured at 37.3℃ for subjects >14 years old and 37.5℃ for subjects <14 years old.
  2. Acute illness or acute onset of chronic disease within 3 days prior to vaccination;
  3. Other conditions for which investigators decide vaccination should be delayed. Exclusion criteria for subsequent dose vaccination:If any of the following occurs during the study safety observation period, subjects may not continue with vaccination, but may continue with other study steps at the discretion of the investigator.

  <!-- -->

  1. Newly discovered or newly occurred before vaccination that did not meet the inclusion criteria (except items with *);
  2. Meet the exclusion criteria for the first dose (except for items with *);
  3. Vaccination-related adverse events occur after vaccination and subsequent doses are not considered appropriate by investigators;
  4. The investigator determines any circumstances that require discontinuation of vaccination from a subject risk and benefit perspective.

Exclusion criteria for immunopersistent blood collection:

1. Incomplete full immunization;
2. Vaccination with rabies immunoglobulin or other rabies vaccines within 12 months after full immunization;
3. Long-term use (>15 days) of immunosuppressants or other immunomodulatory drugs (such as glucocorticoids) within 12 months after full vaccination;
4. Any other circumstances that the investigator believes may affect the evaluation of the trial.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2460 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Antibody SCR in 5-dose groups of test vaccine and 5-dose groups of control vaccine | Day 14
  Antibody Seroconversion rate in 5-dose groups of test vaccine and 5-dose groups of control vaccine
Antibody GMC in 5-dose groups of test vaccine and 5-dose groups of control vaccine | Day 14
  Antibody Geometric Mean Concentration in 5-dose groups of test vaccine and 5-dose groups of control vaccine
Antibody SCR in 4-dose groups of test vaccine and 5-dose groups of control vaccine | Day 14
  Antibody Seroconversion rate in 4-dose groups of test vaccine and 5-dose groups of control vaccine
Antibody GMC in 4-dose groups of test vaccine and 5-dose groups of control vaccine | Day 14
  Antibody Geometric Mean Concentration in 4-dose groups of test vaccine and 5-dose groups of control vaccine
Antibody SCR in 5-dose groups of test vaccine and 5-dose groups of control vaccine | Day 42
  Antibody Seroconversion rate in 5-dose groups of test vaccine and 5-dose groups of control vaccine
Antibody SCR in 4-dose groups of test vaccine and 5-dose groups of control vaccine | Day 42
  Antibody Seroconversion rate in 4-dose groups of test vaccine and 5-dose groups of control vaccine

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Sichuan Center for Disease Control and Prevention, Chengdu, Sichuan
  - Center for Disease Control and Prevention, Mianyang City, Mianyang, Sichuan
  - Shizhong District, Neijiang City Center for Disease Control and Prevention, Neijiang, Sichuan
  - Rongxian Center for Disease Control and Prevention, Zigong, Sichuan